CLINICAL TRIAL: NCT03422107
Title: Clinical Assessment of a Novel Automated SSEP Monitor for Detection and Management of Intraoperative Positional Neuropraxia
Brief Title: Somatosensory Evoked Potential (SSEP) Monitoring for Detection of Intraoperative Positional Neuropraxia
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Western University, Canada (Other)
Responsible Party: Sponsor
Other Study IDs: R-16-286
Record Dates: First submitted 2018-01-29; First posted 2018-02-05 (Actual); Last update posted 2018-03-12 (Actual); Status verified 2018-01

CONDITIONS: Peripheral Nerve Injuries; Thoracic Surgery
Keywords: Peripheral Nerve Injuries; Thoracic Surgery; Minimally invasive cardiac surgery
MeSH Terms: conditions — Peripheral Nerve Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- TAVI: Transcatheter Aortic Valve Implantation
- cAVR: Conventional Valve Replacement
- rCABG: minimally invasive coronary artery bypass graft
- cCABG: Conventional Coronary Artery Bypass Graft

SUMMARY:
PNI (Peripheral Nerve Injury) occurs in 5-15% of patients in cardiac surgery. So far, the mechanism of injury has never been researched. In this study, we will compare minimally invasive cardiac surgery with conventional cardiac surgery using a novel portable SSEP device to pinpoint the mechanism and timing of PNI during cardiac surgery.

DETAILED DESCRIPTION:
General objectives The general objective of this study is to identify the causative insults during various kinds of cardiac surgeries. To attain this objective, we have three specific aims. Firstly, surgical insults such as excessive or asymmetric sternal retraction have long been regarded as the main causes of PNI. Therefore, we will investigate this by comparing cardiac surgeries with sternotomy to the ones without sternotomy. Secondly, more and more cardiac surgeons utilize minimally invasive techniques these days. In the current study, we will investigate the incidence, mechanisms and patterns of PNI in minimally invasive cardiac surgeries by comparing conventional surgeries to minimally invasive surgeries. Thirdly, recent studies have suggested systematic insults such as ischemia, inflammation, and underlying neuropathy might play more prominent roles in the mechanism of PNI. In this study, we will analyze various factors such as intraoperative hemodynamics and baseline patient characteristics to pinpoint the most responsible factors.

Background The studies regarding mechanisms of PNI in cardiac surgeries have not been done over the past few decades. With respect to minimally invasive cardiac surgeries, no studies have been done to investigate the mechanism of PNI.

Regarding the device used in this study The conventional SSEP device is large in size, invasive, and requires expertise to interpret. These characteristics have prevented its use in the operating room. This new portable SSEP device is devoid of these properties.

Significance Identification of causative insults will help clinicians to recognize and possibly prevent PNI during cardiac surgeries.

ELIGIBILITY:
Inclusion Criteria:

●all adult (age>18, <95 years of age) cardiac surgical patients who are undergoing the four following procedures, open AVR, TAVI, conventional CABG, robotic CABG

Exclusion Criteria:

* any patients with contraindication to SSEP monitoring, which include skin burns or trauma at SSEP electrode sites
* lack of written consent
* emergency surgery
* language barrier
* fluctuating neurological signs/symptoms
* regional anesthesia (spinal, epidural, nerve block)
* CABG with radial artery harvest, combined cardiac surgeries

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Our inclusion criteria are all adult (age>18 years of age) cardiac surgical patients who are undergoing the four following procedures, open AVR, TAVI, conventional CABG, robotic CABG. This 4 groups of patients represent 4 different combination of potential surgical insults- median sternotomy, Internal thoracic artery (ITA) retraction, ITA harvesting, cardiopulmonary bypass and positioning
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2017-11-20 (Actual); Primary Completion 2018-12-31 (Estimated); Study Completion 2019-06-30 (Estimated)

PRIMARY OUTCOMES:
Cumulative duration of abnormal SSEP | From the beginning of the surgery to the end of surgery
  Defined as the amplitude reduction >50% from baseline, Latency>10% from baseline

SECONDARY OUTCOMES:
The incidence of postoperative peripheral neuropathy at post-operative day 2-5 | Post operative day 2 to 5
  The incidence of postoperative peripheral neuropathy at Post-operative day (POD) 2-5, which is diagnosed based on neurological examination
The number of SSEP abnormal alarms | From the beginning of the surgery to the end of surgery
  The frequencies the SSEP devise sets off alarms

CONTACTS AND LOCATIONS:
Overall Officials: John Murkin, MD, Study Director — Western University
Locations (1):
- London Health Sciences Centre, London, Ontario, Canada